CLINICAL TRIAL: NCT00025168
Title: Phase II Trial Of Induction Gemcitabine/CPT-11 Followed By Twice-Weekly Infusion Gemcitabine And Concurrent External Beam Radiation For The Treatment Of Locally Advanced Pancreatic Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Locally Advanced Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: REBACDR0000068933; CCCWFU-57100; NCI-5332
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Irinotecan; Radiotherapy

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: irinotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and irinotecan, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and radiation therapy in treating patients who have locally advanced, unresectable pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the time to progression, local control, and survival of patients with locally advanced, unresectable pancreatic cancer treated with induction gemcitabine and irinotecan followed by gemcitabine and concurrent radiotherapy.

OUTLINE: Patients receive induction gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1 and 8. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Within 2 weeks of completing induction chemotherapy, patients receive gemcitabine IV over 30-60 minutes on days 1, 4, 8, 11, 15, 18, 22, 25, 29, and 32. Patients undergo concurrent radiotherapy 5 days a week for 5.5 weeks.

Patients are followed every 8 weeks for 6 months and then every 3 months for 1.5 years.

PROJECTED ACCRUAL: Approximately 60-120 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced pancreatic cancer
* Regional (peri-pancreatic) lymph node involvement allowed
* Clinically or surgically staged and considered unresectable or inoperable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 6 months

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Hemoglobin at least 10 g/dL
* Platelet count at least 100,000/mm3

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant
* Fertile patients must use effective contraception
* No other concurrent or prior malignancy within the past 2 years except nonmelanoma skin cancer or in situ carcinoma of the cervix or breast
* No other serious medical or psychiatric illness that would preclude giving informed consent or limit survival to less than 2 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent anticancer immunotherapy

Chemotherapy:

* No prior chemotherapy
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent anticancer hormonal therapy

Radiotherapy:

* No prior abdominal-pelvic radiotherapy
* No other concurrent anticancer radiotherapy

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior open abdominal surgery
* More than 10 days since prior laparoscopy

Other:

* No other concurrent investigational drug
* No concurrent participation in other clinical study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-11-01 (Actual); Primary Completion 2003-08-29 (Actual); Study Completion 2003-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur William Blackstock, MD, Study Chair — Wake Forest University Health Sciences
Locations (7):
- United States (7):
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina

REFERENCES:
- [Result] Mishra G, Butler J, Ho C, Melin S, Case LD, Ennever PR, Magrinat GC, Bearden JD, Minotto DC, Howerton R, Levine E, Blackstock AW. Phase II trial of induction gemcitabine/CPT-11 followed by a twice-weekly infusion of gemcitabine and concurrent external beam radiation for the treatment of locally advanced pancreatic cancer. Am J Clin Oncol. 2005 Aug;28(4):345-50. doi: 10.1097/01.coc.0000159559.42311.c5. PMID 16062075